CLINICAL TRIAL: NCT02820441
Title: Adaptative Servoventilation Compliance in Left Ventricular Dysfunction Patients With Central Sleep Apnea: Benefit of One Month Hypnotic (Zopiclone) Versus Placebo
Brief Title: Benefit of One Month Zopiclone Intake on Adaptative Servoventilation Compliance
Acronym: ZODIAC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 38RC15.175
Record Dates: First submitted 2016-06-07; First posted 2016-07-01 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2016-06

CONDITIONS: Sleep Apnea, Central; Ventricular Dysfunction
MeSH Terms: conditions — Sleep Apnea, Central; Ventricular Dysfunction | interventions — zopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZOPICLONE (Experimental): Zopiclone 3.5 mg capsule by mouth daily for 2 weeks
  Interventions: Drug: Zopiclone
- PLACEBO (Placebo Comparator): Placebo 3.5 mg capsule by mouth daily for 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zopiclone
  Other Names: IMOVANE
  Arms: ZOPICLONE
Drug: Placebo
  Arms: PLACEBO

SUMMARY:
The study evaluate the effect of adaptative servoventilation (ASV) initiation combined with 14 days Zopiclone vs Placebo treatment in patients with central sleep apnea (CSA) syndrome.

DETAILED DESCRIPTION:
ASV remain the optimal treatment for CSA in Heart Failure patients with preserved left ventricular ejection fraction (LVEF).

Yet, the adaptation to the ventilation is extremely challenging and the resulting difficulties encountered to sleep induction might be a reason for dropping out.

Zopiclone is indicated for the short-term treatment of insomnia where sleep initiation or sleep maintenance are prominent symptoms. In this study, Zopiclone, as sedative and hypnotic agent, is used during the ASV initiation period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 90 years at the initial visit
* Central Sleep Apnea with an AHI ≥ 15/h and at least 50% of central events indicating an ASV therapy, as determined by a ventilatory polygraphy (PG) or a polysomnography (PSG)
* Cardiac Dysfunction with Left Ventricular Ejection fraction(LVEF)> 45% determined by a transthoracic echocardiography (TTE), known for more than 12 weeks and stable for at least 4 weeks;
* Compliance less than 3 hours after 7 days of the setting up of ASV;
* Patient affiliated to a social security scheme or being beneficiary of such scheme;
* Patient voluntarily participating in the research, with written informed consent

Exclusion Criteria:

* Current use of continuous positive airway pressure (cPAP) for treatment of sleep apnea during the last 12 months
* Presence of chronic symptomatic heart failure with reduced left ventricular ejection fraction (LVEF ≤ 45%), and a CSA moderate to severe (AHI ≥15 / h)
* Presence of severe pulmonary bullous disease
* Presence of Pneumothorax or pneumomediastinum
* Hypotension, especially if associated with depletion of intravascular volume
* Dehydration
* Leaking of cerebrospinal fluid, cranial surgery or trauma recently.
* Episode of acute respiratory failure or heart failure in the previous month

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Average use of the Adapative Servo Ventilation device per day assessed by the device data | one month
  daily use of the device (hours/day, mean value), amount of hours and number of day the device has been used as assessed by the device data

SECONDARY OUTCOMES:
Average use of the Adapative Servo Ventilation device per day assessed by the device data | 3 months and 12 months
Residual Apnea, Hypopnea Index (number/hour) | 12 months
  Index assessed by device data
Daytime sleepiness assessed by the Epworth Sleepiness Scale (ESS) | 1 month
Daytime sleepiness assessed by the Epworth Sleepiness Scale (ESS) | 3 months
Daytime sleepiness assessed by the Epworth Sleepiness Scale (ESS) | 12 month
Asthenia assessed by Pichot scale | 1 month
Asthenia assessed by Pichot scale | 3 months
Asthenia assessed by Pichot scale | 12 months
Changes in New York Heart Association score | 1 month
Changes in New York Heart Association score | 3 months
Changes in New York Heart Association score | 12 months
Number of prescription of hypnotics drug | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie DESTORS, MD, Principal Investigator — University Hospital, Grenoble Alpes, FRANCE
Locations (1):
- Clinique de Physiologie Sommeil et Exercice, Pole Thorax et Vaisseaux , University Hospital Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boccon-Gibod I, Bouillet L. [Angioedema and urticaria]. Ann Dermatol Venereol. 2014 Nov;141 Suppl 3:S586-95. doi: 10.1016/S0151-9638(14)70162-0. French. PMID 25539680
- [Background] Pagnier A. [Hereditary angioedema in childhood. Diagnosis and therapeutic challenges]. Presse Med. 2015 Jan;44(1):89-95. doi: 10.1016/j.lpm.2014.07.018. Epub 2014 Dec 12. French. PMID 25511651
- [Background] Dinkel HP, Maroske J, Schrod L. Sonographic appearances of the abdominal manifestations of hereditary angioedema. Pediatr Radiol. 2001 Apr;31(4):296-8. doi: 10.1007/s002470000409. PMID 11321752
- [Background] Bygum A. Hereditary angio-oedema in Denmark: a nationwide survey. Br J Dermatol. 2009 Nov;161(5):1153-8. doi: 10.1111/j.1365-2133.2009.09366.x. Epub 2009 Jun 22. PMID 19709101
- [Background] Farkas H. Pediatric hereditary angioedema due to C1-inhibitor deficiency. Allergy Asthma Clin Immunol. 2010 Jul 28;6(1):18. doi: 10.1186/1710-1492-6-18. PMID 20667121
- [Background] El-Hachem C, Amiour M, Guillot M, Laurent J. [Hereditary angioneurotic edema: a case report in a 3-year-old child]. Arch Pediatr. 2005 Aug;12(8):1232-6. doi: 10.1016/j.arcped.2005.03.052. French. PMID 15890504
- [Background] Farkas H. Management of upper airway edema caused by hereditary angioedema. Allergy Asthma Clin Immunol. 2010 Jul 28;6(1):19. doi: 10.1186/1710-1492-6-19. PMID 20667122
- [Background] Sanchez A, Ecochard A, Maestracci M, Rodiere M. [Hereditary angioedema causing colocolic intussusception]. Arch Pediatr. 2008 Mar;15(3):271-4. doi: 10.1016/j.arcped.2007.12.004. Epub 2008 Mar 10. French. PMID 18329867
- [Background] Pritzker HA, Levin TL, Weinberg G. Recurrent colocolic intussusception in a child with hereditary angioneurotic edema: reduction by air enema. J Pediatr Surg. 2004 Jul;39(7):1144-6. doi: 10.1016/j.jpedsurg.2004.03.075. PMID 15213920
- [Background] Parisi G, Chiarelli A, Squadrone NP, Galante E. Hereditary angioedema, a rare cause of recurrent abdominal pain. A report of 2 clinical cases and comments of a general nature Allergy Asthma Proc. 2013 Jul-Aug;34(4):312-27
- [Background] MacGinnitie AJ. Pediatric hereditary angioedema. Pediatr Allergy Immunol. 2014 Aug;25(5):420-7. doi: 10.1111/pai.12168. Epub 2013 Dec 9. PMID 24313851
- [Background] Deroux A, Vilgrain I, Dumestre-Perard C, Boccon-Gibod I, Bouillet L. Towards a specific marker for acute bradykinin-mediated angioedema attacks: a literature review. Eur J Dermatol. 2015 Jul-Aug;25(4):290-5. doi: 10.1684/ejd.2015.2547. PMID 25905454
- [Background] Nussberger J, Cugno M, Cicardi M. Bradykinin-mediated angioedema. N Engl J Med. 2002 Aug 22;347(8):621-2. doi: 10.1056/NEJM200208223470820. No abstract available. PMID 12192030
- [Background] Cugno M, Zanichelli A, Bellatorre AG, Griffini S, Cicardi M. Plasma biomarkers of acute attacks in patients with angioedema due to C1-inhibitor deficiency. Allergy. 2009 Feb;64(2):254-7. doi: 10.1111/j.1398-9995.2008.01859.x. Epub 2008 Dec 4. PMID 19076541
- [Background] Hogan AD, Schwartz LB. Markers of mast cell degranulation. Methods. 1997 Sep;13(1):43-52. doi: 10.1006/meth.1997.0494. PMID 9281467
- [Background] Brickman CM, Frank MM, Kaliner M. Urine-histamine levels in patients with hereditary angioedema (HAE). J Allergy Clin Immunol. 1988 Sep;82(3 Pt 1):403-6. doi: 10.1016/0091-6749(88)90012-7. PMID 3170987
- [Background] Payne V, Kam PC. Mast cell tryptase: a review of its physiology and clinical significance. Anaesthesia. 2004 Jul;59(7):695-703. doi: 10.1111/j.1365-2044.2004.03757.x. PMID 15200544
- [Background] Kasperska-Zajac A, Grzanka A, Czecior E, Misiolek M, Rogala B, Machura E. Acute phase inflammatory markers in patients with non-steroidal anti-inflammatory drugs (NSAIDs)-induced acute urticaria/angioedema and after aspirin challenge. J Eur Acad Dermatol Venereol. 2013 Aug;27(8):1048-52. doi: 10.1111/j.1468-3083.2012.04486.x. Epub 2012 Feb 21. PMID 22348297
- [Background] Fujii K, Konishi K, Kanno Y, Ohgou N. Acute urticaria with elevated circulating interleukin-6 is resistant to anti-histamine treatment. J Dermatol. 2001 May;28(5):248-50. doi: 10.1111/j.1346-8138.2001.tb00126.x. PMID 11436361
- [Background] Kasperska-Zajac A, Brzoza Z. Increased D-dimer concentration in plasma of patients with severe acute urticaria. Br J Dermatol. 2009 Dec;161(6):1409-10. doi: 10.1111/j.1365-2133.2009.09466.x. Epub 2009 Sep 15. No abstract available. PMID 19754863
- [Background] Brevet: w/o 2008 062314 circulating ve-cadherin as a predictive marker of sensitivity or resistance to anti-tumoral treatment, and improved method for the detection of soluble proteins.
- [Background] Bouillet L, Sidibe A, Polena H, Mannic T, Deroux A, Stidder B, Vittecoq O, Vilgrain I. [Endothelial junctions: exploiting their instability in the development of biomarkers for vascular remodelling]. Med Sci (Paris). 2014 Jun-Jul;30(6-7):633-5. doi: 10.1051/medsci/20143006012. Epub 2014 Jul 11. No abstract available. French. PMID 25014453
- [Background] Bouillet L, Vilgrain I. VE-cadherin, a potential marker for endothelial cell activation during hereditary angioedema attacks. J Allergy Clin Immunol. 2014 Jul;134(1):241. doi: 10.1016/j.jaci.2014.04.016. Epub 2014 May 27. No abstract available. PMID 24875615
- [Background] Sidibe A, Polena H, Pernet-Gallay K, Razanajatovo J, Mannic T, Chaumontel N, Bama S, Marechal I, Huber P, Gulino-Debrac D, Bouillet L, Vilgrain I. VE-cadherin Y685F knock-in mouse is sensitive to vascular permeability in recurrent angiogenic organs. Am J Physiol Heart Circ Physiol. 2014 Aug 1;307(3):H455-63. doi: 10.1152/ajpheart.00774.2013. Epub 2014 May 23. PMID 24858856
- [Background] Sidibe A, Polena H, Razanajatovo J, Mannic T, Chaumontel N, Bama S, Marechal I, Huber P, Gulino-Debrac D, Bouillet L, Vilgrain I. Dynamic phosphorylation of VE-cadherin Y685 throughout mouse estrous cycle in ovary and uterus. Am J Physiol Heart Circ Physiol. 2014 Aug 1;307(3):H448-54. doi: 10.1152/ajpheart.00773.2013. Epub 2014 May 23. PMID 24858855
- [Background] Bouillet L, Mannic T, Arboleas M, Subileau M, Massot C, Drouet C, Huber P, Vilgrain I. Hereditary angioedema: key role for kallikrein and bradykinin in vascular endothelial-cadherin cleavage and edema formation. J Allergy Clin Immunol. 2011 Jul;128(1):232-4. doi: 10.1016/j.jaci.2011.02.017. Epub 2011 Mar 24. No abstract available. PMID 21439626
- [Background] Suffritti C, Zanichelli A, Maggioni L, Bonanni E, Cugno M, Cicardi M. High-molecular-weight kininogen cleavage correlates with disease states in the bradykinin-mediated angioedema due to hereditary C1-inhibitor deficiency. Clin Exp Allergy. 2014 Dec;44(12):1503-14. doi: 10.1111/cea.12293. PMID 24552232
- [Background] Kahn R, Herwald H, Muller-Esterl W, Schmitt R, Sjogren AC, Truedsson L, Karpman D. Contact-system activation in children with vasculitis. Lancet. 2002 Aug 17;360(9332):535-41. doi: 10.1016/S0140-6736(02)09743-X. PMID 12241658
- [Background] Ghannam A, Sellier P, Defendi F, Favier B, Charignon D, Lopez-Lera A, Lopez-Trascasa M, Ponard D, Drouet C. C1 inhibitor function using contact-phase proteases as target: evaluation of an innovative assay. Allergy. 2015 Sep;70(9):1103-11. doi: 10.1111/all.12657. Epub 2015 Jun 9. PMID 26010015
- [Background] Adam SS, Key NS, Greenberg CS. D-dimer antigen: current concepts and future prospects. Blood. 2009 Mar 26;113(13):2878-87. doi: 10.1182/blood-2008-06-165845. Epub 2008 Nov 13. PMID 19008457
- [Background] Blohme G. Treatment of hereditary angioneurotic oedema with tranexamic acid. A random double-blind cross-over study. Acta Med Scand. 1972 Oct;192(4):293-8. doi: 10.1111/j.0954-6820.1972.tb04818.x. No abstract available. PMID 4562897
- [Background] Brown NJ, Gainer JV, Stein CM, Vaughan DE. Bradykinin stimulates tissue plasminogen activator release in human vasculature. Hypertension. 1999 Jun;33(6):1431-5. doi: 10.1161/01.hyp.33.6.1431. PMID 10373228
- [Background] Cugno M, Hack CE, de Boer JP, Eerenberg AJ, Agostoni A, Cicardi M. Generation of plasmin during acute attacks of hereditary angioedema. J Lab Clin Med. 1993 Jan;121(1):38-43. PMID 8426080
- [Background] Frank MM, Sergent JS, Kane MA, Alling DW. Epsilon aminocaproic acid therapy of hereditary angioneurotic edema. A double-blind study. N Engl J Med. 1972 Apr 13;286(15):808-12. doi: 10.1056/NEJM197204132861503. No abstract available. PMID 4551861
- [Background] Joseph K, Tholanikunnel BG, Wolf B, Bork K, Kaplan AP. Deficiency of plasminogen activator inhibitor 2 in plasma of patients with hereditary angioedema with normal C1 inhibitor levels. J Allergy Clin Immunol. 2016 Jun;137(6):1822-1829.e1. doi: 10.1016/j.jaci.2015.07.041. Epub 2015 Sep 26. PMID 26395818
- [Background] Kaplan AP, Austen KF. A prealbumin activator of prekallikrein. II. Derivation of activators of prekallikrein from active Hageman factor by digestion with plasmin. J Exp Med. 1971 Apr 1;133(4):696-712. doi: 10.1084/jem.133.4.696. PMID 4251126
- [Background] Kleniewski J, Blankenship DT, Cardin AD, Donaldson V. Mechanism of enhanced kinin release from high molecular weight kininogen by plasma kallikrein after its exposure to plasmin. J Lab Clin Med. 1992 Jul;120(1):129-39. PMID 1535355
- [Background] Kluft C, Trumpi-Kalshoven MM, Jie AF, Veldhuyzen-Stolk EC. Factor XII-dependent fibrinolysis: a double function of plasma kallikrein and the occurrence of a previously undescribed factor XII- and kallikrein-dependent plasminogen proactivator. Thromb Haemost. 1979 Jun 30;41(4):756-73. PMID 483248
- [Background] Nielsen EW, Johansen HT, Hogasen K, Wuillemin W, Hack CE, Mollnes TE. Activation of the complement, coagulation, fibrinolytic and kallikrein-kinin systems during attacks of hereditary angioedema. Scand J Immunol. 1996 Aug;44(2):185-92. doi: 10.1046/j.1365-3083.1996.d01-298.x. PMID 8711433
- [Background] Reshef A, Zanichelli A, Longhurst H, Relan A, Hack CE. Elevated D-dimers in attacks of hereditary angioedema are not associated with increased thrombotic risk. Allergy. 2015 May;70(5):506-13. doi: 10.1111/all.12587. Epub 2015 Feb 23. PMID 25640891